CLINICAL TRIAL: NCT04662268
Title: Assessment of a Composite Prognostic Score to Predict Severe Forms of Ischemic Colitis of Montpellier
Brief Title: Assessment of a Composite Prognostic Score to Predict Severe Forms of Ischemic Colitis
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0639
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Ischemic Colitis
Keywords: Ischemic colitis; computed tomography
MeSH Terms: conditions — Colitis, Ischemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our objective is to determine a prognostic score including CT, clinical and biological criteria predicting the serious (death / surgery) or non-serious (medical treatment) evolution of ischemic colitis and therefore possibly modify the therapeutic management (propose surgical treatment for a severe form based on prognostic score).

ELIGIBILITY:
Inclusion criteria:

* Age > or = at 18 years old;
* Performing an abdomino-pelvic scan injected within 6 hours of the onset of symptoms;
* Ischemic colitis proven by endoscopy or surgical data.

Exclusion criteria:

* CT scan performed without injection and / or after 6 hours following the onset of symptoms;
* Unproven ischemic colitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Single-center retrospective cohort (center: CHU de Montpellier) of patients admitted between january 2014 and december 2019 at the CHU, over 18 years of age and having presented ischemic colitis during their stay, with completion of an injected abdomino-pelvic scanner within 6 hours of onset of symptoms, then proven by surgery or endoscopy
Sampling Method: Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Complication rate of ischemic colitis | 1 day
  Severe (surgery and/or death) or non severe form of ischemic colitis (medical treatment) : analysis of radiological, biological and clinical data is performed at the time of acute episode of ischemic colitis when the patient is admitted to the hospital or during the stay of the patient previously present in the hospital for another condition

CONTACTS AND LOCATIONS:
Overall Officials: Patrice TAOUREL, MD-PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC